CLINICAL TRIAL: NCT04771234
Title: Self-guided Digital Psychological Self-care for Individuals With Sleep Problems - Feasibility and Preliminary Effects
Brief Title: Digital Psychological Self-care for Sleep Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Susanna Jernelöv, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-06197
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Insomnia
Keywords: Digital tool; Self-guided
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Pragmatic, within-group pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): The intervention consists of a self-guided digital tool to guide participants with chronic insomnia through sleep restriction and stimulus control procedures.
  Interventions: Behavioral: Digital self-guided CBT-i

INTERVENTIONS:
Behavioral: Digital self-guided CBT-i — A brief version of CBT-i consisting of brief psychoeducation, and the core components sleep restricion and stimulus control, where sleep restriction is based on a simplified sleep diary.
  Other Names: Self-care digital tool

SUMMARY:
In this non-randomized treatment feasibility pilot we want to explore if a simplified version of CBT-i as a non-therapist-guided digital tool can work; if the digital tool is perceived as user friendly and if participants' insomnia severity is improved following four weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia complaints of at least medium severity (15 or above on the ISI)
* Insomnia disorder according to DSM-5
* Adequate language skills (Swedish)
* No foreseeable practical hinders to participate
* Can wear actigraph 24/7
* Daily access to the internet, via computer, smart phone or tablet

Exclusion Criteria:

* Sleep disorders requiring other treatment (e.g. sleep apnea)
* Somatic or psychiatric disorders that require other treatment (e.g. suicide risk, severe depression) or that decrease level of functioning enough to prevent working independently.
* Use of alcohol or drugs in a way that will affect sleep negatively, use of medications with a negative impact on sleep. (Stable use of anti depressants and stable use or tapering of hypnotics are allowed)
* Night work or shift work involving night work
* Ongoing or previous psychological treatment including sleep restricion and stimulus control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | From base-line to 4 weeks
  7-item self-reported measure of insomnia severity, 0-28 Points. Higher values represents higher severity (worse outcome)
Insomnia Severity Index | From base-line to 20 weeks
  7-item self-reported measure of insomnia severity, 0-28 Points. Higher values represent higher severity (worse outcome)
Treatment acceptability/usefulness | From base-line to 4 weeks
  Qualitative quesions regarding participant perception of using the digital tool (ease of use, whether the tool was helpful)

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | From base-line to 4 weeks
  9-item self-report measure of depression severity, 0-28 points. Higher values represent higher severity (worse outcome)
Patient Health Questionnaire (PHQ-9) | From base-line to 20 weeks
  9-item self-report measure of depression severity, 0-28 points. Higher values represent higher severity (worse outcome)
Generalized Anxiety Disorder Scale (GAD7) | From base-line to 4 weeks
  7-item self-report measure of anxiety severity, 0-21 points. Higher values represent higher severity (worse outcome)
Generalized Anxiety Disorder Scale (GAD7) | From base-line to 20 weeks
  7-item self-report measure of anxiety severity, 0-21 points. Higher values represent higher severity (worse outcome)

OTHER OUTCOMES:
Adverse events and Negative effects questionnaire (NEQ) | From base-line to 4 weeks
  Self-report measures of negative effects and adverse events; Higher values represent more adverse events and negative effects
Actigraphy | From base-line to 4 weeks
  A wrist-worn device to measure sleep, giving measures of e.g. total sleep time, wake after sleep onset, and sleep efficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Program for Anxiety and Affective disorders, Stockholm Southwest Psychiatry, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No